CLINICAL TRIAL: NCT04472702
Title: Fluoroscopic Versus Ultrasound Guidance for Cooled Radiofrequency Ablation of Geniculate Nerves in Knee Osteoarthritis: A Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: American Medical Society for Sports Medicine Collaborative Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1868999; STUDY00005460 (Other: University of Rochester)
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants (N=90; 45 at each site) will be randomized with equal probability to either treatment group, restricted by equal enrollment and equal distribution at each site. Patients will be enrolled for the exploratory aim separately at the University of Florida site only. After enrollment into the main study (primary and secondary aims), subjects at the UF site will be offered enrollment into the exploratory aim (N=24) on a consecutive basis restricted by equal enrollment into each treatment arm. A random number table will be used for group allocation and the values recorded separately into opaque, sealed envelopes. This will be performed by a clinical coordinator who is not involved in study to ensure allocation concealment. Outcomes for the primary, secondary, and exploratory aims will be completed by research staff who are blinded to the subject treatment allocation. Data analyses will also be completed in a blinded fashion by the study statistical consultant.
Who Masked: Investigator
Masking Description: A random number table will be used for group allocation and the values recorded separately into opaque, sealed envelopes. This will be performed by a clinical coordinator who is not involved in study to ensure allocation concealment. Outcomes for the primary, secondary, and exploratory aims will be completed by research staff who are blinded to the subject treatment allocation. Data analyses will also be completed in a blinded fashion by the study statistical consultant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Subjects with knee OA using ultrasound for cRFA intervention (Experimental): Knee osteoarthritis patients (Kellegren-Lawrence Scale 2-4) that have been refractory to conservative treatments and report at least 80% pain relief with diagnostic geniculate nerve blocks will be enrolled and randomized to ultrasound (N=45) cRFA treatment arm.
  Interventions: Procedure: cRFA
- Subjects with knee OA using fluoroscopy for cRFA intervention (Experimental): Knee osteoarthritis patients (Kellegren-Lawrence Scale 2-4) that have been refractory to conservative treatments and report at least 80% pain relief with diagnostic geniculate nerve blocks will be enrolled and randomized to fluoroscopic (N=45) cRFA treatment arm.
  Interventions: Procedure: cRFA

INTERVENTIONS:
Procedure: cRFA — cRFA intervention will occur under sterile conditions, the patient will be placed in a supine position on a table and a bolster to provide flexion in the treated knee joint. Skin and soft tissues will be anaesthetized with 2 mL 1% lidocaine at each of the three anatomic sites for cRFA, and a introducer needle will then be placed under ultrasound or fluoroscopic guidance to the SLG, SMG, and IMG nerves. Adjustments at these positions will be made when using ultrasound guidance in order to capture the geniculate nerve if the nerve and/or its accompanying vasculature can be directly visualized using greyscale or Doppler modes. When using ultrasound, the physician will note and record whether their positioning of the needle is based on bony landmarks, direct visualization of the nerve, and/or vascularity accompanying the nerve. Once the introducer needle is placed, the cRFA will be placed into the introducer needle.

SUMMARY:
Cooled radiofrequency ablation (cRFA) of the knee geniculate nerves is a promising treatment option for knee osteoarthritis, but has variable efficacy. Fluoroscopy is the typical guidance of choice, but uses bony landmarks to target these nerves which have variable positions around the knee. Alternatively, ultrasound allows for targeting based on visualization of bony landmarks, the nerves, and their accompanying vascular structures, and thus may offer greater accuracy. However, there are few studies which directly compare the clinical efficacy of these two guidance options. This study will compare these two options.

DETAILED DESCRIPTION:
Background: Cooled radiofrequency ablation (cRFA) of the knee geniculate nerves is a promising treatment option for knee osteoarthritis, but has variable efficacy. Fluoroscopy is the typical guidance of choice, but uses bony landmarks to target these nerves which have variable positions around the knee. Alternatively, ultrasound allows for targeting based on visualization of bony landmarks, the nerves, and their accompanying vascular structures, and thus may offer greater accuracy. However, there are few studies which directly compare the clinical efficacy of these two guidance options. Objective: To compare the effectiveness of geniculate nerve cRFA on knee osteoarthritis outcomes when using either ultrasound or fluoroscopic guidance. The primary outcome measures will be patient pain levels and patient-reported function. The secondary outcome measures will be objective performance-based functional outcomes. The exploratory outcome measures will be blood biomarkers of inflammation, extracellular matrix turnover, and cartilage degradation. Methods: Knee osteoarthritis patients (Kellegren-Lawrence Scale 2-4) that have been refractory to conservative treatments and report at least 80% pain relief with diagnostic geniculate nerve blocks will be enrolled and randomized to fluoroscopic (N=45) or ultrasound (N=45) cRFA treatment arms. Baseline assessments will include 1) Numeric Pain Rating Scale, Western Ontario and McMaster Universities Osteoarthritis Index, and PROMIS depression and pain interference measures; 2) the Osteoarthritis Research Society International recommended physical performance assessments including the 30-Second Chair Stand Test, Stair Climb Test, 40m Fast Paced Walk Test, Timed Up and Go Test, and Six Minute Walk Test; and 3) in a subset of patients (N=24), blood biomarkers including MMP-3, IL-1β, TNF-α, COMP, and CTX-II. These measures will be re-assessed at one month (pain and patient-reported function only, via phone contact), three months, and 6 months after the cRFA procedure. Study endpoints will be assessed using a mixed model repeated measures analysis of variance using an alpha level of 0.05. Statement of Relevance: Knee osteoarthritis patients are commonly treated by sports medicine providers, who are typically well-trained in the use of ultrasound. Should ultrasound be demonstrated as effective for cRFA, sports medicine providers would be well-positioned to use relatively low-cost and accessible imaging technology to significantly improve patient pain and function using cRFA.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients of either gender with primary knee OA of one or both knees fulfilling the diagnostic criteria for knee OA by the American College of Rheumatology,
* 2) Kellgren-Lawrence score of two to four,
* 3) reported NPRS pain intensity of at least four on most or all days of the past week
* 4) pain resistant to conventional treatments which may include but is not limited to medications (e.g. acetaminophen, oral or topical non-steroidal anti-inflammatory drugs, opioids), physical therapy, and intra-articular injections (e.g. corticosteroids, hyaluronic acid, platelet-rich-plasma) for at least 3 months. In the case of bilateral knee OA, the most symptomatic knee will be treated and studied.

Exclusion Criteria:

* 1) age <35 years,
* 2) non-English speaking patients,
* 3) body mass index greater than 40,
* 4) previous radiofrequency ablation procedure for the knee,
* 5) active systemic or local infections at the site of needle/cRFA probe placement,
* 6) previous knee joint replacement surgery,
* 7) autoimmune or inflammatory cause of knee arthritis such as rheumatoid or psoriatic arthritis,
* 8) non-ambulatory patients,
* 9) patients who are unable to provide their own consent (e.g. dementia),
* 10) unstable medical or psychiatric illness,
* 11) patients with pacemakers, spinal cord stimulators, deep brain stimulators, or similar devices,
* 12) patients seeking care as a part of workman's compensation or have litigation pending
* 13) a negative response to diagnostic geniculate nerve lidocaine injections.

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline up to 24 months
  The objective is to rate patient's reported pain. The NPRS asks for a number between zero and ten that fits best to the subject's pain intensity, with zero as "no pain at all" and ten representing "the worst pain ever possible". It has a similar minimal clinically significant difference (20%) as the visual analog scale and can be administered via a phone interview.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline up to 24 months
  The objective is to measure the patient's reported functional status.The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores
PROMIS - Depression | Baseline up to 24 months
  The objective is to measure items relevant to the subject's mood, views of self, and engagement. The test version 8b has good responsiveness with a minimally important difference range of 3-3.1 in adults with knee OA.
PROMIS - Pain Interference | Baseline up to 24 months
  The objective is to measure the consequences of pain on the subject's life with a minimally important difference range of 2.35 to 2.4

SECONDARY OUTCOMES:
30-Second Chair Stand Test | The subjects will perform the OARSI-recommended performance-based functional tests at the baseline, three month, and six month time periods.
  The objective is to determine the maximum number of chair stand repetitions possible in a 30 second period.
Stair Climb Test | The subjects will perform the OARSI-recommended performance-based functional tests at the baseline, three month, and six month time periods.
  The objective is to determine the time (seconds) it takes to ascend and descend a flight of stairs.
40m Fast Paced Walk Test | The subjects will perform the OARSI-recommended performance-based functional tests at the baseline, three month, and six month time periods.
  The objective is to determine the time (seconds) it takes to complete a fast-paced walking task over 4x10m (total 40m).
Timed Up and Go Test48 | The subjects will perform the OARSI-recommended performance-based functional tests at the baseline, three month, and six month time periods.
  The objective is to determine the time (seconds) to rise from a chair, walk 3m, turn, walk back to the chair, and then sit down.
Six Minute Walk Test | The subjects will perform the OARSI-recommended performance-based functional tests at the baseline, three month, and six month time periods.
  The objective is to determine the maximal distance covered in a 6min period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Herman, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UC Davis Health, Sacramento, California
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No